CLINICAL TRIAL: NCT03675802
Title: Randomized Comparison of Vaginal Dinoprostone and Misoprostol for Cervical Ripening Before Diagnostic Hysteroscopy in Patients Who Have Undergone Cesarean Section
Brief Title: Cervical Preparation in Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Hysteroscopy
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female | interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm number one ,misoprostol (Active Comparator)
  Interventions: Drug: misoprostol
- Arm number 2 dinoprostone (Active Comparator)
  Interventions: Drug: dinoprostone

INTERVENTIONS:
Drug: misoprostol — giving misoprostol to this group
  Arms: Arm number one ,misoprostol
Drug: dinoprostone — giving dinoprostine
  Arms: Arm number 2 dinoprostone

SUMMARY:
The hysteroscopy was performed in the proliferativephase of the menstrual cycle.

The patients were given generalintravenous anesthesia (propofol/fentanyl) after the vulvar and the vaginal area had been disinfected with a 7.5% Betadinesolution by the surgical nurse All operations were performed by the same surgeon to avoid possible discrepancies between different surgeons.

DETAILED DESCRIPTION:
Astandard rigid30 hysteroscope (Karl Storz bettocchi hysteroscope) with a 30° viewing angleand an outer sheath diameter 5.5 mm, inner sheath diameter 4.3 mm and scope diameter 2.9 mmwas used in all procedures.

A speculum was introduced into the vagina, and the uterine cervixwas visualized. Initially, the surgeon attempted to passthrough the cervical canal with the tool directly. When thatwas not possible or when the cervical canal was too rigid ortoo tight, the cervix was grasped with a tenaculum.

ELIGIBILITY:
Inclusion Criteria:

1. patients of reproductive age
2. have undergone a cesarean section at least once
3. an indication for diagnostic hysteroscopy for menstrualproblems or suspected intrauterine lesions (suchas uterine polyps and ﬁlling defects in the uterine cavity) by abnormal ﬁndings from hysterosalpingography,ultrasonography, or saline infusion sonography.

Exclusion Criteria:

1. Patients who delivered vaginally
2. Had undergone any other transcervical or transabdominal uterine and cervical intervention other than cesareansection, such as loop electrosurgical procedures, cervical cryotherapy, cervical biopsies, and spontaneousabortions, previous dilation, and previous electiveabortions.
3. Patients with cervical pathology,e.g. tears or polyps.
4. The patients with a contraindicationto prostaglandins such as hypersensitivity, bronchial asthma, glaucoma, severeasthma, cardiac, liver or kidney diseases.

   -

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who needs diagnostic hysteroscopy
Enrollment: 100 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
The number of women who will require cervical dilatation | within an hour

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud Alalfy, PhD, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No